CLINICAL TRIAL: NCT03057444
Title: Influence of Resistant Starch Type III on Butyrate-producing Gut Bacteria and Diabetes Parameter in (Pre-) Diabetes
Brief Title: Resistant Starch, Gut Bacteria and Diabetes
Acronym: RSDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Collaborators: Institut für Mikroökologie GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UniHohMet-RSIII-2016
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus, Type 2; Pre Diabetes
Keywords: resistant starch type III; butyrate-producing gut bacteria; diabetes mellitus type 2; prediabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Prediabetic State

STUDY DESIGN:
Intervention Model Description: open intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): The patients get 2x 5g per day the food supplement SymbioIntest (resistant starch types III) over 8 weeks.
  Study examinations are before intervention, after 4 weeks and 8 weeks. Stool samples are collected before intervention and each 14 days consecutively until the end of intervention.
  Interventions: Dietary Supplement: SymbioIntest

INTERVENTIONS:
Dietary Supplement: SymbioIntest — The intervention is 2x 5g per day the food supplement SymbioIntest (resistant starch types III) over 8 weeks.

SUMMARY:
The aim of the study is to investigate, if resistant starch type III increases butyrate-producing bacteria in the gut of (pre-) diabetic subjects. Diabetic blood parameters are also of interest.

DETAILED DESCRIPTION:
Other studies show that diabetics have less butyrate-producing bacteria species in the gut compared to non-diabetes patients and diabetes patients who are taking metformin. Moreover, studies demonstrate that resistant starch increases the butyrate-producing bacteria species. Furthermore, studies show that butyrate has on effect on blood glucose and insulin homeostasis.

The aim in this study is to investigate, if resistant starch typ III increases butyrate-producing bacteria in the gut of (pre-) diabetic subjects, The effects on blood glucose, insulin and HbA1c are investigated as well.

Patients included in the study are typ 2 diabetics with lifestyle interventions, insulin or antidiabetic medication (sulfonylureas, glinides, SGLT2-inhibitors, glitazone) or pre-diabetics.

They get 2x 5g per day the food supplement SymbioIntest (resistant starch types III) over 8 weeks.

Study examinations are before intervention, after 4 weeks and 8 weeks. Stool samples are collected before intervention and each 14 days consecutively until the end of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult persons (≥ 18 years)
* Type 2 diabetes mellitus discontinued with lifestyle interventions or insulin therapy or oral antidiabetic therapy (sulphonylureas, glinides, SGLT-2 (sodium/glucose cotransporter 2) inhibitors, glitazone) or a prediabetic metabolism
* It is foreseeable that no therapy with metformin or α-glucosidase inhibitors or DPP-4 (Dipeptidyl peptidase-4) inhibitors is initiated during the period of study (8 weeks)
* willingness not to systematically change diet and lifestyle habits during the study
* Adequate understanding of the German language and sufficient psychological condition to understand the information and instructions associated with the study and to complete questionnaires and assessment scales
* Signed informed consent

Exclusion Criteria:

* Treatment of Type II diabetes mellitus by metformin or α-glucosidase inhibitors or DPP-4 inhibitors
* Diminished diabetic metabolic position or medical necessity to convert the therapy in the foreseeable future (HbA1c ≥ 7% or fasting glucose ≥ 152 mg / dl)
* Participation in another clinical trial (currently or within the last 30 days)
* Incompatibility with the ingredients of the investigational medicinal product
* Pregnancy or lactation
* Inability to take the test preparation orally
* changes in dietary habits and habits within the last 30 days
* Antibiotics intake currently or within the last 30 days
* Drug abuse in the last six months before the start of the study or ongoing. Alcohol abuse is defined as an average daily of more than 20 g of alcohol in women and more than 30 g of alcohol in men, based on the last six months
* A state of health (including abnormal laboratory values) that, at the discretion of the investigator, does not allow study participation, evaluation of study parameters or the use of the investigational medicinal product
* Accommodation in a clinic or similar facility, by administrative or judicial order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Change of gut bacteria | Participants will be followed for the time of eight weeks. Examinations take place at baseline, four and eight week
  quantitative Analyse with Next-Generation Sequencing
Change of short chain fatty acid concentration in the gut | Participants will be followed for the time of eight weeks. Examinations take place at baseline, four and eight week
  gas chromatography

SECONDARY OUTCOMES:
change from baseline in HbA1c at four weeks and eight weeks after consumption resistant starch type III | Participants will be followed for the time of eight weeks. Examinations take place at baseline, four and eight week.
change from baseline in insulin at four weeks and eight weeks after consumption resistant starch type III | Participants will be followed for the time of eight weeks. Examinations take place at baseline, four and eight week.
change from baseline in blood glucose at four weeks and eight weeks after consumption resistant starch type III | Participants will be followed for the time of eight weeks. Examinations take place at baseline, four and eight week
Change from baseline in anthropometry at four weeks and eight weeks after consumption resistant starch type III | Participants will be followed for the time of eight weeks. Examinations take place at baseline, four and eight week

OTHER OUTCOMES:
Change from baseline in PYY (Peptide YY) at four weeks and eight weeks after consumption resistant starch type III | Participants will be followed for the time of eight weeks. Examinations take place at baseline, four and eight week.
  with ELISA
Change from baseline in GLP-1 (Glucagon-like peptide-1) at four weeks and eight weeks after consumption resistant starch type III | Participants will be followed for the time of eight weeks. Examinations take place at baseline, four and eight week.
  with ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Stephan C. Bischoff, Prof., Principal Investigator — University of Hohenheim, 70599 Stuttgart
Locations (1):
- Institute of Clinical Nutrition, Stuttgart, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No